CLINICAL TRIAL: NCT07016841
Title: Effects of Conventional Hemodialysis Combined With pHA Hemoperfusion Therapy on Protein-Bound Uremic Toxins in Maintenance Hemodialysis Patients: A Single-Center, Prospective Cohort Study
Brief Title: Effects of pHA Hemoperfusion Plus Hemodialysis on Protein-Bound Uremic Toxins
Status: Recruiting | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-25-005
Record Dates: First submitted 2025-05-26; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2024-12

CONDITIONS: End Stage Renal Disease on Dialysis
Keywords: Hemoadsorption; Hemodialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- experimental group: Treatment regimen: Hemodialysis (HD)/Hemodiafiltration (HDF) combined with Hemoperfusion (HP) using the pHA130 hemoperfusion device, with HD administered twice weekly, HDF once weekly (each session lasting 4 hours), and HP once every 2 weeks.
  Interventions: Device: pHA130 hemoperfusion device; Device: HD/HDF
- control group 1: Control Group 1: HD/HDF Treatment regimen: HD twice weekly, HDF once weekly, with each session lasting 4 hours.
  Interventions: Device: HD/HDF
- control group 2: Control Group 2: HD/HDF combined with HP (HA130 hemoperfusion device) Treatment regimen: HD twice weekly, HDF once weekly (each session lasting 4 hours), and HP once every 2 weeks.
  Interventions: Device: HD/HDF; Device: HA130 hemoperfusion device

INTERVENTIONS:
Device: pHA130 hemoperfusion device — HP once every 2 weeks.
  Groups: experimental group
Device: HD/HDF — HD twice weekly, HDF once weekly, with each session lasting 4 hours.
Device: HA130 hemoperfusion device — HP once every 2 weeks.
  Groups: control group 2

SUMMARY:
This single-center, prospective cohort Study evaluates whether adding the pHA130 hemoperfusion cartridge to conventional hemodialysis (HD) or hemodiafiltration (HDF) more effectively reduces protein-bound uremic toxins-specifically indoxyl sulfate (IS) and p-cresyl sulfate (PCS)-in maintenance HD patients. Adults on thrice-weekly, 4-hour HD for at least three months are randomized to one of three arms: HD/HDF alone; HD/HDF plus biweekly pHA130 hemoperfusion; or HD/HDF plus biweekly HA130 hemoperfusion. After a four-week washout, toxin levels are measured at baseline and again at Weeks 4, 12, and 24, with the primary endpoint being the reduction in IS and PCS at Week 24. Secondary endpoints include single-session toxin removal, middle-molecule clearance (β₂-microglobulin, PTH), patient-reported outcomes (itching, sleep, quality of life), and rates of hospitalization and mortality. Safety is closely monitored through adverse event reporting and consistent anticoagulation dosing. Findings will clarify the clinical value of pHA130 hemoperfusion for improving toxin clearance and guiding optimal dialysis strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, with no restriction on gender;
2. Undergoing regular hemodialysis 3 times per week, 4 hours per session, and has received maintenance hemodialysis treatment for ≥3 months;
3. Willing and able to receive treatment as per the protocol requirements, and has signed the informed consent form for subjects.

Exclusion Criteria:

1. Patients receiving combined hemodialysis (HD) and peritoneal dialysis (PD) treatment;
2. Patients with known allergy to hemoperfusion device materials, contraindications, or intolerance to the device;
3. Patients with acute severe infection, severe cardiopulmonary insufficiency, severe cerebrovascular disease, severe bleeding tendency, or active bleeding;
4. Patients with malignant tumors in the active stage or undergoing treatment for malignant tumors;
5. Patients with a platelet count < 60 × 10⁹/L;
6. Other conditions deemed unsuitable for enrollment in this study by the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable maintenance hemodialysis patients meeting the inclusion and exclusion criteria with a dialysis vintage ≥3 months.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Serum indoxyl sulfate (IS) | Week 0 to Week 24 (±7 days)
  value at 24 weeks minus value at baseline reported
Serum p-cresyl sulfate (PCS) | Week 0 to Week 24 (±7 days)
  value at 24 weeks minus value at baseline reported

SECONDARY OUTCOMES:
Parathyroid hormone (PTH) | before/after a single treatment session
  Reduction rate of parathyroid hormone (PTH) before/after a single treatment session
β2-microglobulin (β2-MG) | before/after a single treatment session
  Reduction rate of β2-microglobulin (β2-MG) before/after a single treatment session.
Serum indoxyl sulfate (IS) | before/after a single treatment session
  Reduction rate of serum indoxyl sulfate (IS) before/after a single treatment session
Serum p-cresyl sulfate (PCS) | before/after a single treatment session
  Reduction rate of serum p-cresyl sulfate (PCS) before/after a single treatment session.
Kidney Disease Quality of Life Short Form (KDQOL-SF) Total Score | Week 0 to Week 24 (±7 days)
  Change in KDQOL-SF (Kidney Disease Quality of Life Short Form) total score from baseline to week 24.
Pruritus severity score | Week 0 to Week 24 (±7 days)
  Change from baseline in pruritus severity score (VAS and Modified Duo Pruritus Score) at Week 24.
Pittsburgh Sleep Quality Index (PSQI) | Week 0 to Week 24 (±7 days)
  Change in Pittsburgh Sleep Quality Index (PSQI) from baseline to Week 24
Hospitalization rate | Week 0 to Week 24 (±7 days)
  24-week hospitalization rate (All-cause, cardiovascular event, infection, vascular access event-related and β2-MG-related symptom hospitalization rate)
Mortality rate | Week 0 to Week 24 (±7 days)
  24-week-mortality (All-cause, cardiovascular event, infection, vascular access event-related and β2-MG-related symptom )

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China